CLINICAL TRIAL: NCT07014852
Title: Integrating Inuit Knowledge Principles in Multi-Level Mental Health Clinical Trials
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Aqqiumavvik - Arviat Wellness Society (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Pro00149001
Record Dates: First submitted 2025-05-12; First posted 2025-06-11 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Depression, Anxiety
Keywords: Inuit; Country Foods; mental health; depression; anxiety; food sovereignty; cultural identity; community wellness; Indigenous health; Inuit Qaujimajatuqangit (IQ); social cohesion
MeSH Terms: conditions — Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Intervention (Other): Weekly distributions of traditional country foods (caribou, seal, Arctic char), Elder-led workshops on food preparation and cultural practices, and mental health supports through unnikkaaratiginniq and sharing circles for the first 30 days of the trial.
  Interventions: Other: Traditional Country Foods; Behavioral: Cultural Workshops
- Delayed Intervention (Other): Participating in baseline assessments only (no guided conversations or workshops from Days 1-30). From Days 30-60, the delayed intervention group will receive the same intervention as the immediate intervention group
  Interventions: Other: Traditional Country Foods; Behavioral: Cultural Workshops

INTERVENTIONS:
Other: Traditional Country Foods — Participants will receive weekly distributions of traditional foods, including caribou and fish. Guided conversations will explore changes in dietary habits, emotional well-being, and cultural connections
Behavioral: Cultural Workshops — Weekly workshops led by Elders will focus on traditional country food, food preparation, and sharing practices, enhancing cultural identity and community bonds. Participants will also engage in cultural camps where they will be led by Elders in land based teachings on country food.

SUMMARY:
This study is looking at how eating more country foods affects mental health among Inuit men and women in Arviat, NU. The goal is to evaluate if eating more of these foods helps people feel less depressed or anxious, and whether being part of food-gathering and cultural activities also makes a difference.

Whether the positive effects last over time, and if getting access to these foods later (instead of right away) still helps people feel better, will also be assessed.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the feasibility, cultural acceptability, and potential mental health impacts, measured using PHQ-9 as part of a multi-level intervention (MLI) that integrates country foods, community wellness practices, and clinical care.

Specifically, the intervention aims to:

Improve mental health outcomes: Increased access to country foods is hypothesized to reduce depression and anxiety.

Strengthen cultural identity: Community-led wellness activities are expected to enhance cultural identity and community cohesion.

Enhance food sovereignty: Addressing systemic barriers can improve access to country foods and support culturally relevant healthcare.

Promote continuity of care: Integrating culturally grounded interventions into care plans can improve patient outcomes and overall wellness.

Secondary objectives include assessing the role of Elders in transferring cultural knowledge, identifying systemic barriers to accessing country food, and evaluating the integration of IQ principles into clinical systems. Elders are expected to facilitate social cohesion and transfer cultural knowledge, which are vital for community resilience. Policy recommendations will be explored to address systemic barriers, while the intervention's findings will inform clinical care plans to promote culturally relevant healthcare.

Ultimately, this research aims to develop community-based, culturally aligned solutions that promote resilience, improve health outcomes, and support Inuit self-determination. This study aims to create sustainable pathways for wellness and food sovereignty in Inuit communities by addressing historical injustices and systemic inequities.

Research Question(s): This study is guided by the following research questions:

How does increased access to country foods influence individual mental health outcomes, including anxiety, depression, emotional well-being, and resilience? How do community-driven food-gathering activities enhance social cohesion, cultural identity, and collective mental health within Inuit communities? What structural, systemic, and environmental barriers restrict access to Inuit country foods, and what specific policy interventions can effectively address these barriers to promote sustainable food security and mental health improvements? How do land-based and country food wellness programs integrate holistic approaches to address biological, psychological, social, and cultural determinants of mental health? What role do interdisciplinary collaborations and culturally relevant care practices play in improving access to country foods and fostering mental health equity in Inuit communities?

Hypotheses:

Increased access to country foods will improve mental health outcomes, including reduced depression and anxiety.

Community-led wellness activities will strengthen cultural identity, social bonds, and cohesion.

Access to country foods will help address systemic barriers and enhance food sovereignty while supporting culturally relevant healthcare.

Integrating culturally grounded interventions into care plans will improve continuity of care and patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Inuit
* Able to consent to study participation
* Participating in community wellness programs facilitated by the Aqqiumavvik Wellness Centre within 6 months prior to screening
* Willing to consume country foods provided as part of the intervention
* Willing to engage in individual and group activities, including guided conversations and cultural workshops
* 18-65 years of age

Exclusion Criteria:

* Less than 18 years of age
* Greater than 65 years of age
* Unable to consent to study participation
* Mental health conditions requiring immediate clinical intervention
* Known allergies or medical conditions that prevent the consumption of traditional country foods
* Physical or logistical barriers that prevent participation in weekly activities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2026-09-13 (Estimated); Study Completion 2026-09-20 (Estimated)

PRIMARY OUTCOMES:
Cultural Acceptability of the Intervention- Qualitative Interviews | From enrolment to the end of treatment at 12 weeks
  Qualitative interviews with healthcare providers and community facilitators will explore barriers and facilitators to intervention implementation.
Cultural Acceptability of the Intervention- Participant Diaries | From enrolment to the end of treatment at 12 weeks
  Participant diaries will also be used to assess the perceived cultural significance of the intervention.
Participant satisfaction and perceived impact on mental health | From enrolment to the end of treatment at weeks 4, 8, and 12.
  Data will also be collected through participant diaries, focusing on experiences with country food consumption, the perceived cultural significance of the intervention, and overall satisfaction with the program. REDCap surveys will collect data from participant diaries, allowing for consistent monitoring of cultural experiences and satisfaction over time.
Mental Health Impacts | Baseline (enrolment)
  Potential mental health impacts will be measured using the Patient Health Questionnaire-9 (PHQ-9) tool at baseline. Scoring ranges from 0-27; a higher score indicates worse mental health.
Mental Health Impacts - 4 weeks | 4 weeks after enrolment
  Potential mental health impacts will be measured using the Patient Health Questionnaire-9 (PHQ-9) tool 4 weeks after enrolment. Scoring ranges from 0-27; a higher score indicates worse mental health
Mental Health Impacts | 8 weeks after enrolment
  Potential mental health impacts will be measured using the Patient Health Questionnaire-9 (PHQ-9) tool 8 weeks after enrolment. Scoring ranges from 0-27; a higher score indicates worse mental health.
Mental Health Impacts | 12 weeks after enrolment
  Potential mental health impacts will be measured using the Patient Health Questionnaire (PHQ-9) tool 12 weeks after enrolment. Scoring ranges from 0-27; a higher score indicates worse mental health.
Participant Satisfaction- Participant Diaries | Baseline (at enrolment)
  Data will be collected through participant diaries that focus on experiences with country food consumption, the perceived cultural significance of the intervention, and overall satisfaction with the program at baseline.
Participant Satisfaction- Participant Diaries | 4 weeks after enrolment
  Data will be collected through participant diaries that focus on experiences with country food consumption, the perceived cultural significance of the intervention, and overall satisfaction with the program 4 weeks after enrolment
Participant Satisfaction- Participant Diaries | 8 weeks after enrolment
  Data will be collected through participant diaries that focus on experiences with country food consumption, the perceived cultural significance of the intervention, and overall satisfaction with the program 8 weeks after enrolment
Participant Satisfaction- Participant Diaries | 12 weeks after enrolment
  Data will be collected through participant diaries that focus on experiences with country food consumption, the perceived cultural significance of the intervention, and overall satisfaction with the program 12 weeks after enrolment

SECONDARY OUTCOMES:
Assessment of the Role of Elders in Transferring Cultural Knowledge- Workshops | 12 weeks after enrolment
  Assessment of the Role of Elders in Transferring Cultural Knowledge will be evaluated through Elder-led workshops.
Assessment of the Role of Elders in Transferring Cultural Knowledge- Conversations | 12 weeks after enrolment
  Assessment of the Role of Elders in Transferring Cultural Knowledge will be evaluated through guided unikkaaqatiginniq conversations.
Systemic Barriers to Accessing Country Food- Interviews | 12 weeks after enrolment
  Evaluation of systemic barriers to accessing country food will be done via interviews with health care providers who provide care to Inuit within the region.
Systemic Barriers to Accessing Country Food- Participant Diaries | 12 weeks after enrolment
  Evaluation of systemic barriers to accessing country food will be done via qualitative analysis of participant diaries.
Systemic Barriers to Accessing Country Food- Discussions | 12 weeks after enrolment
  Evaluation of systemic barriers to accessing country food will be done via insights from Circle discussions with participants.
Integration of IQ principles into clinical systems- Participant Diaries | Once between 12-24 weeks after enrolment
  Evaluation of the integration of IQ principles into clinical systems will be done via qualitative analysis of participant diaries. Recommendations will be made to the Government of Nunavut and the Nunavut Health Authority based on this analysis into how IQ principles can be incorporated across the health care and clinical systems.
Integration of IQ principles into clinical systems- Discussions | Once between 12-24 weeks after enrolment
  Evaluation of the integration of IQ principles into clinical systems will be done via insights from Circle discussions with participants. Recommendations will be made to the Government of Nunavut and the Nunavut Health Authority based on this analysis into how IQ principles can be incorporated across the health care and clinical systems.
Integration of IQ principles into clinical systems- Interviews | Once between 12-24 weeks after enrolment
  Evaluation of the integration of IQ principles into clinical systems will be done via interviews with health care providers who provide care to Inuit within the region. Recommendations will be made to the Government of Nunavut and the Nunavut Health Authority based on this analysis into how IQ principles can be incorporated across the health care and clinical systems.

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Clark, Ed.D, Principal Investigator — University of Alberta; Justin Ezekowitz, MD, Principal Investigator — University of Alberta
Locations (2):
- Canada (2):
  - Aqqiumavvik Society, Arviat, Nunavut
  - Aqqiumavvik - Arviat Wellness Society, Arviat, Nunavut

IPD SHARING:
Plan to Share IPD: No
Given the size of the study population, IPD will not be shared.

REFERENCES:
- [Background] Young, T. K. (2012). Health and disease in the Canadian North. University of Toronto Press.
- [Background] Willows ND. Determinants of healthy eating in Aboriginal peoples in Canada: the current state of knowledge and research gaps. Can J Public Health. 2005 Jul-Aug;96 Suppl 3:S32-6, S36-41. English, French. PMID 16042162
- [Background] Wilson, S. (2008). Research is ceremony: Indigenous research methods. Fernwood Publishing.
- [Background] Turner, N. J., Ignace, M. B., & Ignace, R. (2013). Traditional ecological knowledge and wisdom of Aboriginal Peoples in British Columbia. Ecological Applications, 10(5), 1275-1287.
- [Background] Tagalik, S. (2011). Inuit Qaujimajatuqangit: The role of Indigenous knowledge in supporting wellness in Inuit communities. National Collaborating Centre for Aboriginal Health. https://www.nccih.ca/docs/context/FS-InuitQaujimajatuqangitWellness-EN.pdf
- [Background] Austin S. Decolonizing methodologies: research and indigenous people. J Health Psychol. 2001 May;6(3):358-9. doi: 10.1177/135910530100600310. No abstract available. PMID 22049381
- [Background] Santos Dunn, C., Yazzie, M., & Tsosie, R. (2023). Colonial legacies, food sovereignty, and health inequities among Indigenous peoples. Indigenous Policy Journal, 34(1), 1-18.
- [Background] Rink, E. (2019). Intergenerational trauma and resilience among Indigenous youth: A multi-level intervention model. Journal of Adolescent Health, 65(6), 782-789. https://doi.org/10.1016/j.jadohealth.2019.07.014
- [Background] Richmond C, Elliott SJ, Matthews R, Elliott B. The political ecology of health: perceptions of environment, economy, health and well-being among 'Namgis First Nation. Health Place. 2005 Dec;11(4):349-65. doi: 10.1016/j.healthplace.2004.04.003. PMID 15886143
- [Background] Power EM. Conceptualizing food security or aboriginal people in Canada. Can J Public Health. 2008 Mar-Apr;99(2):95-7. doi: 10.1007/BF03405452. PMID 18457280
- [Background] Marmot M. Social justice, epidemiology and health inequalities. Eur J Epidemiol. 2017 Jul;32(7):537-546. doi: 10.1007/s10654-017-0286-3. Epub 2017 Aug 3. PMID 28776115
- [Background] Louis, R. P. (2007). Can you hear us now? Voices from the margin: Using Indigenous methodologies in geographic research. Geographical Research, 45(2), 130-139. https://doi.org/10.1111/j.1745-5871.2007.00443.x
- [Background] LaLonde, C. E., Richmond, C. A., & McGregor, D. (2023). Food security, cultural continuity, and Indigenous health in Canada: The critical role of community initiatives. Canadian Journal of Public Health, 114(1), 45-54. https://doi.org/10.17269/s41997-022-00669-0
- [Background] Kovach, M. (2009). Indigenous methodologies: Characteristics, conversations, and contexts. University of Toronto Press.
- [Background] Kazdin, A. E. (2021). Research design in clinical psychology (5th ed.). Cambridge University Press.
- [Background] Tester FJ, McNicoll P. 'Why don't they get it?' Talk of medicine as science. St Luke's Hospital, Panniqtuuq, Baffin Island. Soc Hist Med. 2006 Apr;19(1):87-106. doi: 10.1093/shm/hkj006. PMID 17153162
- [Background] Healey Akearok, G., Tagalik, S., & Healey, J. (2024). Integrating Inuit Qaujimajatuqangit in clinical trials: A decolonizing approach to mental health research. Canadian Indigenous Health Review, 4(1), 32-50.
- [Background] Healey Akearok, G., Tagalik, S., & Healey, J. (2019). Inuit knowledge and its role in health promotion: Lessons from Nunavut for community-based interventions. Arctic, 72(3), 273-285. https://doi.org/10.14430/arctic69064
- [Background] First Nations Information Governance Centre. (2014). Ownership, Control, Access and Possession (OCAP®): The path to First Nations information governance. First Nations Information Governance Centre.
- [Background] Egeland GM, Johnson-Down L, Cao ZR, Sheikh N, Weiler H. Food insecurity and nutrition transition combine to affect nutrient intakes in Canadian arctic communities. J Nutr. 2011 Sep;141(9):1746-53. doi: 10.3945/jn.111.139006. Epub 2011 Jul 13. PMID 21753059
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] Andrée, P., Dibden, J., Higgins, V., & Cocklin, C. (Eds.). (2023). Globalization and food sovereignty: Global and local change in the new politics of food. Routledge.
- [Background] Baumgartner, R. N. (2024). Multi-level interventions in Indigenous health: Prioritizing systemic change in clinical research funding. Journal of Indigenous Health Research, 9(2), 87-103.
- [Background] Blue Bird Jernigan, V. (2020). Multi-level and community-based interventions for Indigenous populations: Challenges and opportunities. Current Epidemiology Reports, 7(2), 84-91. https://doi.org/10.1007/s40471-020-00233-4
- [Background] Anderson LM, Petticrew M, Rehfuess E, Armstrong R, Ueffing E, Baker P, Francis D, Tugwell P. Using logic models to capture complexity in systematic reviews. Res Synth Methods. 2011 Mar;2(1):33-42. doi: 10.1002/jrsm.32. Epub 2011 Jun 10. PMID 26061598